CLINICAL TRIAL: NCT01222104
Title: Clinical Registry of St. Jude Medical Angio-Seal™ Vascular Closure Devices Following Interventional Radiology Procedures
Brief Title: Angio-Seal Interventional Radiology (IR) Registry
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: 0903
Record Dates: First submitted 2010-10-05; First posted 2010-10-18 (Estimated); Results first posted 2014-11-19 (Estimated); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Diagnostic and/or Interventional Radiology Procedures
Keywords: vascular closure; Angio-Seal; Interventional radiology; femoral artery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Angio-Seal: Angio-Seal attempted and/or deployed
- Not deployed: Other method of closure

SUMMARY:
The purpose of this study is to collect data on the standard of care use of the St. Jude Medical (SJM) Angio Seal™ Evolution™ and V-Twist Integrated Platform (VIP) Devices in diagnostic and/or interventional radiology patient populations.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is undergoing a diagnostic and/or interventional radiology procedure via femoral arterial access and the investigator performing the procedure would use Angio-Seal for closure as part of his/her routine care of the patient. Angio-Seal deployment will follow the standard of care for vascular closure device use and the Instructions for Use (IFU) for the device.
2. Sheath angiography prior to Angio-Seal deployment reveals appropriate anatomy and puncture location for vascular closure device deployment.

Exclusion Criteria:

1. Patients who are unable to provide written informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who undergo a diagnostic and/or interventional radiology procedure through percutaneous femoral artery access and meet the registry selection criteria.
Sampling Method: Probability Sample
Enrollment: 634 (Actual)
Dates: Start 2010-10; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zoltan Turi, M.D., Principal Investigator — Cooper University
Locations (10):
- United States (10):
  - Loma Linda University Medical Center, Loma Linda, California
  - Yale New Haven Hospital, New Haven, Connecticut
  - University of Florida, Gainesville, Florida
  - Baptist Cardiac and Vascular Institute, Miami, Florida
  - University of Kansas Medical Center, Kansas City, Kansas
  - Kaleida Health, Buffalo, New York
  - Mayfield Clinic, Inc.; The University Hospital, Cincinnati, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Thomas Jefferson Hospital, Philadelphia, Pennsylvania
  - Albert Einstein Medical Center, Philadelphia, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | All Participants
Started | 634
Angio-Seal Deployment Attempted | 534
Successful Deployment | 529
Successful Deployment and Hemostasis | 524
Completed 30-day Visit-Angio-Seal | 497
Completed 30-day Visit-No Angio-Seal | 90
Completed | 587
Not Completed | 47
Not completed — Lost to Follow-up | 37
Not completed — Death | 10

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 634
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.6 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 328
  Male | 306
Region of Enrollment [Number; unit: participants]
  United States | 634

OUTCOME MEASURES:

1. Primary Outcome: Rate of Major Vascular Complications
Description: Collect data on patients who have undergone a diagnostic and/or interventional radiology procedure in which the St. Jude Medical (SJM) Angio-Seal Evolution or V-Twist Integrated Platform (VIP) Device was deployed, to evaluate the rate of major vascular complications out to 30 days post-procedure.
  The following are defined as a major vascular complication:
  1. Vascular injury requiring repair via surgery, angioplasty, ultrasound guided compression, thrombin injection, or other means;
  2. Permanent (unresolved at 30-day post-procedure evaluation) access site-related nerve injury or access site-related nerve injury requiring intervention;
  3. Access site related bleeding requiring transfusion;
  4. New ipsilateral lower extremity ischemia requiring surgical intervention;
  5. Retroperitoneal bleeding;
  6. Generalized infection requiring prolonged hospitalization and/or treatment with IV antibiotics;
  7. Access related complication that results in extended hospital stay;
  8. Death
Time Frame: 30 days
Population: 5 subjects underwent vascular closure with Angio-Seal on right and left sides.
Measure: Number; unit: Percentage of Procedures
Units Other Than Participants: Procedures
Groups:
- Angio -Seal: Angio-Seal attempted and/or deployed group
Arm/Group | Angio -Seal
Number analyzed (Participants) | 534
Number analyzed (Procedures) | 539
Percentage of Procedures | 0.7

2. Secondary Outcome: Time to Hemostasis
Description: Time-to-hemostasis stratified into 3 categories: hemostasis in less than 1 minute alone or in combination with manual compression (standard of care), 1-5 minutes alone or in combination with manual compression (standard of care), and/or hemostasis achieved >5 minutes and/or with additional hemostasis methods required.
Time Frame: Procedure
Measure: Number; unit: % of procedures
Units Other Than Participants: Procedures
Groups:
- Angio-Seal: Secondary outcome reported in subjects with successful Angio-Seal deployment which achieved hemostasis by device.
Arm/Group | Angio-Seal
Number analyzed (Participants) | 524
Number analyzed (Procedures) | 529
% of procedures
  Hemostasis less than 1 minute | 84.9
  Hemostasis between 1-5 minutes | 13.0
  Hemostasis greater than 5 minutes | 2.1

3. Secondary Outcome: Rate of Minor Vascular Complications
Description: The following are defined as a minor vascular complication:
  1. Unanticipated access site bleeding requiring ≥ 30 minutes of manual compression to re-achieve hemostasis;
  2. Ipsilateral hematoma >10 cm;
  3. Ipsilateral pseudoaneurysm without intervention;
  4. Ipsilateral arteriovenous fistula;
  5. Ipsilateral deep vein thrombosis;
  6. Local access site infection without prolonged hospitalization
Time Frame: 30 days
Measure: Number; unit: % of procedures with minor vasc comp.
Units Other Than Participants: Procedures
Arm/Group | All Participants
Number analyzed (Participants) | 534
Number analyzed (Procedures) | 539
% of procedures with minor vasc comp. | 0.7

4. Secondary Outcome: Impact of Guided Access on Use of Closure Device.
Description: The influence of fluoroscopy and/or ultrasound guided access on the decision to use a closure device.
Time Frame: 30 days
Population: Percentage of procedures with devices deployed
Measure: Number; unit: % of procedures using a closure device
Units Other Than Participants: Procedures
Groups:
- All Participants: All enrolled participants
Arm/Group | All Participants
Number analyzed (Participants) | 634
Number analyzed (Procedures) | 639
% of procedures using a closure device
  Ultrasound only, n=30 procedures | 90.0
  Fluorscopy only, n=309 procedures | 86.7
  Fluoro and ultrasound, n=144 procedures | 88.2
  Neither fluoro nor ultrasound, n=156 procedures | 73.1

5. Secondary Outcome: Impact of Guided Access on Achieving Target Puncture Location.
Description: The influence of fluoroscopy and/or ultrasound guided access on puncture location.
Time Frame: 30 days
Population: Deployed subjects with readable angiograms
Measure: Number; unit: % within target zone
Arm/Group | All Participants With Deployments and Readable Angiograms
Number analyzed (Participants) | 468
% within target zone
  Ultrasound only, n=23 participants | 87.0
  Fluoroscopy only, n=240 participants | 81.7
  Both Fluoro and ultrasound, n=113 participants | 77.0
  Neither fluoro nor ultrasound, n=92 participants | 87.0

6. Secondary Outcome: Rate of Major Vascular Complications (MVCs) by Guided Access Mode.
Description: The influence of fluoroscopy and/or ultrasound guided access on Major Vascular Complications (MVCs).
Time Frame: 30 days
Measure: Number; unit: % of procedures with MVCs
Units Other Than Participants: Procedures
Groups:
- Participants With Deployments: Participants with successful or attempted Angio-Seal deployments
Arm/Group | Participants With Deployments
Number analyzed (Participants) | 534
Number analyzed (Procedures) | 539
% of procedures with MVCs
  Ultrasound only, n=27 procedures | 0
  Fluoroscopy only, n=269 procedures | 1.1
  Fluoro and ultrasound, n=128 procedures | 0.8
  Neither fluoro nor ultrasound, n=115 procedures | 0

7. Secondary Outcome: Rate of Minor Vascular Complications by Guided Access Mode.
Description: The influence of fluoroscopy and/or ultrasound guided access on minor vascular complications.
Time Frame: 30 days
Measure: Number; unit: % of procedures with minor vasc comp.
Units Other Than Participants: Procedures
Arm/Group | Participants With Deployments
Number analyzed (Participants) | 534
Number analyzed (Procedures) | 539
% of procedures with minor vasc comp.
  Ultrasound only, n=27 procedures | 0
  Fluoroscopy only, n=269 procedures | 0.7
  Fluoro and ultrasound, n=128 procedures | 1.6
  Neither fluoro nor ultrasound, n=115 procedures | 0

8. Secondary Outcome: Impact of Peripheral Vascular Disease (PVD) on Use of Closure Device
Description: Presence of peripheral vascular disease (PVD) and its effect on the decision to use a closure device
Time Frame: 30 days
Measure: Number; unit: % of procedures using closure device
Units Other Than Participants: Procedures
Arm/Group | All Participants
Number analyzed (Participants) | 634
Number analyzed (Procedures) | 639
% of procedures using closure device
  Non-PVD procedures, n=248 | 93.1
  PVD procedures, n=391 | 78.0

9. Secondary Outcome: Impact of Peripheral Vascular Disease (PVD) on Achieving Hemostasis by Device
Description: Presence of peripheral vascular disease (PVD) and its effect on hemostasis. Initial hemostasis by device achieved.
Time Frame: 30 days
Measure: Number; unit: % of procedures achieving hemostasis
Units Other Than Participants: Procedures
Arm/Group | Participants With Deployments
Number analyzed (Participants) | 534
Number analyzed (Procedures) | 539
% of procedures achieving hemostasis
  Non-PVD procedures, n=232 | 98.7
  PVD procedures, n=307 | 97.7

10. Secondary Outcome: Rate of Major Vascular Complications (MVC) by Presence of Peripheral Vascular Disease (PVD)
Description: Presence of peripheral vascular disease (PVD) and its effect on Major Vascular Complications (MVC).
Time Frame: 30 days
Measure: Number; unit: % of procedures with MVCs
Units Other Than Participants: Procedures
Arm/Group | Participants With Deployments
Number analyzed (Participants) | 534
Number analyzed (Procedures) | 539
% of procedures with MVCs
  Non-PVD procedures, n=232 | 0.4
  PVD procedures, n=307 | 1

11. Secondary Outcome: Rate of Minor Vascular Complications by Presence of Peripheral Vascular Disease (PVD)
Description: Presence of peripheral vascular disease (PVD) and its effect on minor vascular complications.
Time Frame: 30 days
Measure: Number; unit: % of procedures with minor vasc comp.
Units Other Than Participants: Procedures
Groups:
- Participants With Deployment: Participants with successful or attempted Angio-Seal deployments
Arm/Group | Participants With Deployment
Number analyzed (Participants) | 534
Number analyzed (Procedures) | 539
% of procedures with minor vasc comp.
  Non-PVD procedures, n=232 | 1.3
  PVD procedures, n=307 | 0.3

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 15/634
Other Adverse Events (participants affected / at risk) | 4/634
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=634)
Vascular injury requiring repair via surgery or other means (Vascular disorders) | 2
New ipsilateral lower extremity ischemia requiring intervention (Vascular disorders) | 1
Retroperitoneal bleeding (Gastrointestinal disorders) | 2
Death (General disorders) | 10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=634)
Ipsilateral hematoma >10cm (Vascular disorders) | 4

LIMITATIONS AND CAVEATS:
Major and minor vascular complications were collected as Serious Adverse Event and Other Adverse Events as defined in the protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days